CLINICAL TRIAL: NCT01859793
Title: A Randomized, Crossover Design Study of Acute and Chronic Effects of Sitagliptin on Endothelial Function in Humans With Type 2 Diabetes on Background Metformin
Brief Title: Effects of Sitagliptin on Endothelial Function in Type 2 Diabetes on Background Metformin Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Michael E. Widlansky, Associate Professor of Medicine, Medical College of Wisconsin
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Merck-50600
Record Dates: First submitted 2013-05-17; First posted 2013-05-22 (Estimated); Results first posted 2016-10-21 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-08

CONDITIONS: Diabetes; Atherosclerosis
Keywords: dipeptidyl peptidase-4 inhibitor; endothelium, vascular; diabetes type 2; nitric oxide; inflammation
MeSH Terms: conditions — Diabetes Mellitus; Atherosclerosis; Diabetes Mellitus, Type 2; Inflammation | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Matching Placebo (Placebo Comparator): Matching Placebo for Sitagliptin
  Interventions: Drug: Placebo
- Sitagliptin (Active Comparator): 100mg pill, PO administered once daily.
  Interventions: Drug: sitagliptin

INTERVENTIONS:
Drug: sitagliptin — 100 mg pill, administered once/day orally
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Placebo — Matching placebo in appearance given once/day orally
  Arms: Matching Placebo

SUMMARY:
The study is being performed to determine whether sitagliptin, a dipeptidyl peptidase-4 inhibitor, both acutely and chronically improves blood vessel function. Patients with type 2 diabetes who are on metformin will be enrolled in this study for up to 22 weeks in this double blinded cross over study where they will receive a sitagliptin pill once a day for 8 weeks and during a separate 8 weeks receive a matching placebo pill. The treatment periods are divided by a 4 week period. Blood vessel function will be measured by ultrasound before and after a single dose of sitagliptin and placebo, as well as after 8 weeks of treatment with each. Blood will also be taken to measure blood markers of inflammation at each time the ultrasounds are performed.

DETAILED DESCRIPTION:
We plan to recruit 38 patients with T2DM for this single center, double blind randomized, interventional crossover trial comparing sitagliptin (100 mg/day) to matching placebo. We have chosen placebo over a comparator for this study as our goal is to determine whether sitagliptin both improves glycemic control and endothelial function, properties not shared by other popular classes of agents like sulfonylureas. Subjects will be randomized with a 1:1 allocation ratio to either sitagliptin 1st or placebo 1st.

The study have 5 total visits. Subjects who pass a phone screen will be invited to a screening visit for study eligibility (Visit 1) Informed consent will be reviewed; a unique study number will be assigned once written informed consent is obtained (no subject will be assigned more than 1 allocation number); relevant participant medical history will be recorded including currently prescribed medications; anthropometric measurements will be taken (height, weight, and waist circumference in metric units) and blood pressure will be recorded (measured in triplicate and averaged). Subjects will be allowed to take their blood pressure medication on the morning of their screening visit, but not the mornings of any of the other study visits to limit the acute influence of these medications on endothelial function. If the potential participant qualifies for the study, he/she will be randomized either to receive sitagliptin 1st (100 mg/day) or matching placebo. Prior to receiving either of set of pills, subjects will return to the study center within approximately 1-2 weeks of the screening visit to undergo initial tests of endothelial function and receive their pills. Prior to all study visits except screening, subjects will also be asked to refrain from any vigorous physical activity (no weight lifting, jogging or any activity vigorous than walking) 24 hours to reduce the risk of fasting hypoglycemia during the study visits. Subjects will also be asked to fast for 6-8 hours prior to the visit to limit the acute dietary influences on vascular endothelial function. At Visit 2, endothelial function will determined by brachial artery reactivity testing prior to and following a single dose of 100 mg of sitagliptin or matching placebo depending on the arm to which the subject was randomized. Blood samples will also be taken at this visit for systemic measurements of endothelial cell activation/inflammation (VCAM-1 and ICAM-1) prior to and 2 hours following acute drug administration. These will be measured at the indicated time points using commercially available kits.

Endothelial function, like the blood samples, will be measured just prior to medication administration and then 2 hours following medication administration by brachial artery reactivity testing as described in Section D.3. The 2 hour time from was chose in given the plasma levels of sitagliptin appear to peak 2 hours following dose administration.32 At the end of this visit, subjects will be given a 9 week supply of the study pills (sitagliptin or matching placebo) as dispensed by the Froedtert Hospital Investigational Pharmacy, and scheduled to return for Visit 3 approximately 8 weeks following Visit 2. Subjects will be asked to not take any study medication for the 24 hours prior to Visit 3. At Visit 3, subjects will undergo repeat testing of endothelial function. Following this study visit, subjects will remain off study pills until they return for Visit 4 approximately 4 weeks following Visit 3. Visit 4 repeats Visit 2 except subjects will receive the set of pills to which they had been randomized to receive second. Subjects will return to the study center for Visit 5 approximately 8 weeks after Visit 4. Visit 5 is identical to Visit 3. Subject adherence will be determined by pill counts performed by MCW Translational Research Unit nursing staff who will perform all pill accounting. All medication dispensation will be handled by the Froedtert Hospital Investigational Drug Pharmacy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult age 21-70 years of age.
2. Diagnosis of type 2 diabetes by a physician as defined by the American Diabetes Association standard criteria: 1) Fasting Plasma glucose at or above 126 mg/dL 2) a two-hour value in an oral glucose tolerance test at or above 200 mg/dL, or 3) a random plasma glucose concentration 200 mg/dL in the presence of symptoms, or 4) glycosylated hemoglobin greater than or equal to 6.5%.
3. On stable metformin therapy for at least 6 weeks prior to enrollment.
4. Glycosylated Hemoglobin ≥6.2% and ≤ 9.5%.

Exclusion Criteria:

1. History of stroke, peripheral arterial disease, or coronary artery disease (as defined by the presence of at least one coronary stenosis ≥ 50% on angiography or by confirmed history of myocardial infarction by standard criteria.)
2. Evidence of other evident major illness including chronic renal insufficiency (creatinine clearance less than 60 mL/min),chronic liver disease (AST or ALT greater than 2.5 x normal), or cancer currently undergoing systemic therapy or had systemic therapy for cancer within 1 year of enrollment.
3. Pregnancy as determined by urinary beta-HCG test
4. Illicit drug use (heroin, cocaine etc) in the past 1 year.
5. Alcohol abuse, defined as the equivalent of 14 beers/week for a man or 7 beers/week for a woman
6. History of allergy to DPP-4 inhibitors at the time of screening/enrollment
7. Prior history of pancreatitis
8. Patients currently on insulin or sulfonylurea therapy.
9. Patients currently on digoxin.

   -

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-06; Primary Completion 2016-01 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael E Widlansky, MD, MPH, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Data set may be shared in a de-identified manner by request from qualified investigators with appropriate qualifications

REFERENCES:
- [Derived] Widlansky ME, Puppala VK, Suboc TM, Malik M, Branum A, Signorelli K, Wang J, Ying R, Tanner MJ, Tyagi S. Impact of DPP-4 inhibition on acute and chronic endothelial function in humans with type 2 diabetes on background metformin therapy. Vasc Med. 2017 Jun;22(3):189-196. doi: 10.1177/1358863X16681486. Epub 2017 Feb 1. PMID 28145158

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo 1st Then Sitagliptin: Matching Placebo for Sitagliptin
  Placebo: Matching placebo in appearance given once/day orally for 8 weeks followed by 8 weeks of 100 mg sitaglipin/day separated by a 4 week washout period
- Sitagliptin First Then Placebo: sitagliptin: 100 mg pill, administered once/day orally for 8 weeks followed by matching placebo for 8 weeks following a 4 week washout period.
Period: First Intervention (8 Weeks)
Arm/Group | Placebo 1st Then Sitagliptin | Sitagliptin First Then Placebo
Started | 20 | 18
Completed | 15 | 17
Not Completed | 5 | 1
Not completed — Protocol Violation | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1
Period: Washout Period (4 Weeks)
Arm/Group | Placebo 1st Then Sitagliptin | Sitagliptin First Then Placebo
Started | 15 | 17
Completed | 14 | 16
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1
Period: 2nd Intervention Period
Arm/Group | Placebo 1st Then Sitagliptin | Sitagliptin First Then Placebo
Started | 14 | 16
Completed | 14 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Matching Placebo 1st: Matching Placebo for Sitagliptin
  Placebo: Matching placebo in appearance given once/day orally
- Sitagliptin 1st: 100mg pill, PO administered once daily.
  sitagliptin: 100 mg pill, administered once/day orally
- Total: Total of all reporting groups
Arm/Group | Matching Placebo 1st | Sitagliptin 1st | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (10) | 63 (9) | 63 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 10 | 14
  Male | 10 | 6 | 16
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 10 | 15 | 25
  Non-Caucasian | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 14 | 16 | 30
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 32.1 (6.6) | 32.6 (6.3) | 32.4 (6.3)
HgA1C [Mean (Standard Deviation); unit: percent] | 6.8 (0.2) | 6.9 (0.8) | 6.8 (0.6)
Heart Rate [Mean (Standard Deviation); unit: bpm] | 72 (10) | 76 (8) | 74 (11)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 131 (13) | 136 (15) | 134 (14)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 73 (11) | 78 (20) | 75 (8)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 165 (31) | 169 (29) | 167 (30)
High Density Lipoprotein [Mean (Standard Deviation); unit: mg/dL] | 55 (12) | 56 (20) | 55 (16)
Low Density Lipoprotein [Mean (Standard Deviation); unit: mg/dL] | 85 (29) | 84 (26) | 84 (27)
Triglycerides [Mean (Standard Deviation); unit: mg/dL] | 126 (53) | 138 (40) | 132 (46)
Insulin [Mean (Standard Deviation); unit: microU/mL] | 15.1 (5.6) | 16.0 (8.9) | 15.6 (7.4)
Glucose [Mean (Standard Deviation); unit: mg/dL] | 117 (26) | 134 (31) | 126 (30)
Homeostatic Assessment of Insulin Resistance [Mean (Standard Deviation); unit: units on a scale] | 4.4 (1.9) | 5.3 (2.9) | 4.9 (2.5)
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: mg/dL] | 30 (30) | 28 (23) | 29 (26)
Aspartate Aminotransferase (AST) [Mean (Standard Deviation); unit: mg/dL] | 25 (17) | 25 (13) | 25 (15)
Total Bilirubin [Mean (Standard Deviation); unit: mg/dL] | 0.4 (0.2) | 0.5 (0.3) | 0.5 (0.3)
Alkaline Phosphatase [Mean (Standard Deviation); unit: mg/dL] | 73 (10) | 78 (20) | 78 (16)
History of Hypertension [Number; unit: participants]
  With Hypertension | 10 | 10 | 20
  Without Hypertension | 4 | 6 | 10
History of High Cholesterol [Number; unit: participants]
  With Dyslipidemia | 8 | 13 | 21
  Without Dyslipidemia | 6 | 3 | 9
Smoking Status [Number; unit: participants]
  Never | 9 | 13 | 22
  Past or Current | 5 | 3 | 8
ACE Inhibitor [Number; unit: participants]
  Yes | 10 | 8 | 18
  No | 4 | 8 | 12
Beta-Blocker [Number; unit: participants]
  Yes | 1 | 1 | 2
  No | 13 | 15 | 28
HMG CoA-Reductase [Number; unit: participants]
  Yes | 9 | 13 | 22
  No | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Brachial Artery Flow Mediated Dilation
Description: A measurement of endothelial function in humans
Time Frame: Change before and after a single dose (2 hours post) and 8 weeks after daily dosing
Population: All 30 subjects who completed both arms of the cross-over study
Measure: Mean (Standard Deviation); unit: %FMD
Arm/Group | Matching Placebo | Sitagliptin
Number analyzed (Participants) | 30 | 30
%FMD
  Prior To Intervention | 5.2 (1.8) | 5.6 (2.3)
  2 hours post acute dose | 5.6 (2.1) | 6.3 (2.4)
  Following 8 weeks of therapy | 6.0 (2.9) | 5.8 (2.3)
Statistical Analysis 1: Comparison: Matching Placebo vs Sitagliptin; Primary and secondary outcome variables were compared across measurement periods by repeated measures ANOVA and post hoc analyses using Tukey's test were applied if significant differences were detected. A priori sample size calculation demonstrated our study design has 80% power to detect a 1.5% absolute increase in FMD% with 30 subjects completing the entire study protocol at α=0.05; Test type: Superiority or Other; p < 0.05, ANOVA

2. Secondary Outcome: Circulating Inflammatory Marker ICAM-1
Time Frame: Change before and after acute dose (2 hours) and 8 weeks after daily dosing of medication
Population: 29 of the 30 subjects who completed both arms of the study. One subject was missing the measurements post 8 weeks of each intervention arm and was excluded
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Matching Placebo | Sitagliptin
Number analyzed (Participants) | 29 | 29
mg/mL
  Pre-Intervention | 226 (72) | 223 (73)
  2 hours post acute dose | 216 (73) | 211 (68)
  post 8 weeks of therapy | 228 (73) | 232 (74)
Statistical Analysis 1: Comparison: Matching Placebo vs Sitagliptin; Outcome variables were compared across measurement periods by repeated measures ANOVA and post hoc analyses using Tukey's test were applied if significant differences were detected; Test type: Superiority or Other; p < 0.05, ANOVA

3. Secondary Outcome: Circulating Inflammatory Markers VCAM-1
Time Frame: Change before and after acute dose (2 hours) and 8 weeks after daily dosing of medication
Population: 29 of the 30 subject who completed the study. Once subject had missing data for the post-8 weeks of each intervention
Measure: Mean (Standard Deviation); unit: mg/mL
Arm/Group | Matching Placebo | Sitagliptin
Number analyzed (Participants) | 29 | 29
mg/mL
  Pre-Intervention | 584 (187) | 608 (164)
  2 hours post acute dose | 575 (141) | 574 (157)
  post 8 weeks of therapy | 620 (196) | 620 (196)
Statistical Analysis 1: Comparison: Matching Placebo vs Sitagliptin; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Matching Placebo | Sitagliptin
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/32
Other Adverse Events (participants affected / at risk) | 1/36 | 0/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Matching Placebo (N=36) | Sitagliptin (N=32)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — 1 subject developed a minor rash along the subjects belt line during the study and was withdrawn from the study. The subject was on placebo at the time as discovered following unblinding

LIMITATIONS AND CAVEATS:
No limitations noted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No